CLINICAL TRIAL: NCT03830021
Title: Effect of a Multi-component Education Program on Salt Reduction in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Cuf Descobertas (Network)
Collaborators: CUF Academic and Research Medical Center (Unknown); José de Mello Saúde (Unknown); Pingo Doce (Unknown); NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ReEducSal001
Record Dates: First submitted 2019-01-28; First posted 2019-02-05 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt reduction program (Experimental): Salt reduction program.
  Interventions: Behavioral: Salt reduction program
- Healthy lifestyle program (Active Comparator): Healthy lifestyle program.
  Interventions: Behavioral: Healthy lifestyle program

INTERVENTIONS:
Behavioral: Salt reduction program — Dietary and behavioural change program, led by nutritionists, including low sodium dietary advice; use of aromatic herbs and spices in food instead of salt; motivational activities; food diaries; restrict salty processed foods; eat more fresh foods and seasoning advice; problem solving exercises; digital bulletins; individual counselling reinforced at each clinic visit and shopping counselling at local supermarket.
  Arms: Salt reduction program
Behavioral: Healthy lifestyle program — Participants receive an educational healthy lifestyle program that includes 1) methods to cook healthier and the Mediterranean diet based on a high intake of fresh fruit and, vegetables, beans, grain legumes, lentils, nuts, cereals, and olive oil as source of fat; moderate intake of fish, poultry, yoghurt and cheese, low intake of salt, red meat, processed meats and sugar; 2) physical activity; 3) drink more water and reducing alcohol consumption; and 4) sleep education.
  Arms: Healthy lifestyle program

SUMMARY:
Excess salt intake is a major contributor to high blood pressure, the leading individual risk factor for cardiovascular events, such as stroke, myocardial infarction and heart failure. According to PHYSA study, salt intake in Portugal remains much higher (10.7 g) than recommended by the international health organisations, indicating the need for effective implementation of salt reduction interventions. In Portugal the main source of daily salt intake is added salt during cooking, and salt content in bread, cheese and processed meat.

The objective of this study is to determine the effectiveness of a dietary education program tailored for salt reduction. To assess the effectiveness of the salt reduction program the investigator's will measure changes in salt consumption levels, by evaluating the 24 h urinary sodium excretion.

This study is a consortium-initiated, randomised, simple-blinded, controlled trial designed to assess the effectiveness of a salt reduction program versus generic healthy lifestyle program in the Lisbon Metropolitan Area.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 20 and 70.
* Subjects with or without hypertension, not medicated or medicated with medication and diet stabilized for at least 3 weeks.
* Responsible for the purchase and confection of their meals.
* Available to comply with study protocol and sign informed consent.

Exclusion Criteria:

* Pregnant, breastfeeding or planning to become pregnant within the study period.
* Subjects with current or previous cardiovascular disease (ischemic cardiovascular disease, angina stable or unstable; myocardial infarction, stroke or symptomatic peripheral arteriosclerosis).
* Subjects with liver or kidney diseases or cancer.
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to cooperate during the study.
* Subjects with special dietary needs.
* Health condition that prevents compliance with study requirements.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urinary sodium excretion | 12 weeks
  Difference between the intervention and control group in the change in 24-hour urinary sodium excretion from baseline to the end of follow-up.

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure | 12 week
  Difference between the intervention and control group in the change in systolic and diastolic blood pressure from baseline to the end of follow-up.
Change in weight | 12 week
  Difference between the intervention and control group in the change of weight from baseline to the end of follow-up.
Change in waist circumference | 12 week
  Difference between the intervention and control group in the change of waist circumference from baseline to the end of follow-up.
Change in salt content in foods purchased | 12 weeks
  Difference between the intervention and control group in the change of salt content in foods purchased from baseline to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Polónia, PhD, Principal Investigator — CINTESIS, Faculty of Medicine of the University of Porto; Conceição Calhau, PhD, Principal Investigator — NOVA Medical School
Locations (2):
- Portugal (2):
  - Hospital CUF Infante Santo, Lisbon
  - Hospital CUF Descobertas, Lisbon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polonia J, Martins L, Pinto F, Nazare J. Prevalence, awareness, treatment and control of hypertension and salt intake in Portugal: changes over a decade. The PHYSA study. J Hypertens. 2014 Jun;32(6):1211-21. doi: 10.1097/HJH.0000000000000162. PMID 24675681
- [Background] Polonia J, Monteiro J, Almeida J, Silva JA, Bertoquini S. High salt intake is associated with a higher risk of cardiovascular events: a 7.2-year evaluation of a cohort of hypertensive patients. Blood Press Monit. 2016 Oct;21(5):301-6. doi: 10.1097/MBP.0000000000000205. PMID 27495189
- [Background] Polonia J, Lobo MF, Martins L, Pinto F, Nazare J. Estimation of populational 24-h urinary sodium and potassium excretion from spot urine samples: evaluation of four formulas in a large national representative population. J Hypertens. 2017 Mar;35(3):477-486. doi: 10.1097/HJH.0000000000001180. PMID 27898506
- [Derived] Moreira-Rosario A, Ismael S, Barreiros-Mota I, Morais J, Rodrigues C, Castela I, Mendes IC, Soares MI, da Costa LS, Oliveira CB, Henriques T, Pinto P, Pita D, de Oliveira CM, Maciel J, Serafim T, Araujo J, Rocha JC, Pestana D, Silvestre MP, Marques C, Faria A, Polonia J, Calhau C. Empowerment-based nutrition interventions on blood pressure: a randomized comparative effectiveness trial. Front Public Health. 2023 Nov 13;11:1277355. doi: 10.3389/fpubh.2023.1277355. eCollection 2023. PMID 38026295